CLINICAL TRIAL: NCT04130165
Title: Optimizing the Prebiotic Profile of Donor Human Milk for Preterm Infants: Feasibility of a New Donor Milk Matching Strategy Based on Maternal Secretor Status
Brief Title: Matching Donor Human Milk On Maternal Secretor Status (MMOMSS) Study
Acronym: MMOMSS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: A variety of feasibility issues.
Sponsor: University of Manitoba (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Meghan Azad, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB19-0542
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Microbial Colonization; Preterm Birth
Keywords: preterm infants; human milk; microbiome; donor human milk; breastmilk
MeSH Terms: conditions — Communicable Diseases; Premature Birth

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor (lab technician/research assistant) will not be aware of the group allocation or nutritional intake of the infant while completing data analysis.
  We cannot blind participants or care providers as provision of matched donor human milk will require preparation which deviates from standard protocol, and the bedside nurse will need to conduct this preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matched donor human milk (Experimental): Infants randomized to the matched donor human milk arm, will receive donor human milk which is matched to their mother's secretor status.
  Interventions: Other: Matched donor human milk
- Standard issue donor human milk (No Intervention): Infants randomized to the standard issue donor human milk arm, will receive donor human milk which is prepared without consideration of secretor status as per standard practice.

INTERVENTIONS:
Other: Matched donor human milk — Milk from donor mothers will be sorted according to their secretor status. This milk will be provided to infants in the intervention (experimental) arm.
  Arms: Matched donor human milk

SUMMARY:
This study will evaluate the impact of matching donor human milk to the maternal secretor status of very preterm infants (<34 weeks gestation) on the gut microbiome. Half of enrolled infants will receive donor human milk which is matched their mother's secretor status and half will receive standard (unmatched) donor human milk, which is standard care in the neonatal intensive care unit.

DETAILED DESCRIPTION:
Background: The gut microbiome is established early in life and plays an important role in developing the immune system and metabolism. Infants born prematurely (before 37-weeks gestation) account for 1 in 10 births worldwide and are especially vulnerable to serious microbiome-mediated illnesses such as necrotizing enterocolitis and metabolic diseases. Breastfeeding is the most important factor shaping the infant gut microbiome, providing human milk oligosaccharides (HMOs) that serve as prebiotics for beneficial gut bacteria. Donor human milk (DHM) is considered the best alternative when mothers own milk (MOM) is not available. HMO profiles are highly variable between mothers and there is currently no "matching" process to optimize pairing of DHM and recipient infants. The strongest factor influencing HMO composition is maternal secretor status, determined by the expression of a specific gene (α-1, 2-fucosyltransferase-2). About 20% of Caucasians are non-secretors and researchers do not know the impact of feeding DHM from secretor donors to infants of non-secretor mothers. In this study, investigators aim to explore if matching DHM based on maternal secretor status impacts the development of the gut microbiome in preterm infants.

Method: Investigators will use a pilot, randomized, controlled trial to compare three groups of preterm infants (<34 weeks gestation): 1) infants receiving DHM matched to their mother's secretor status, 2) infants receiving standard issue (i.e. unmatched) DHM, and 3) infants who do not require DHM because they are exclusively receiving MOM. Mothers <34 weeks gestation admitted to antenatal units and the labour and delivery units will be screened for eligibility. Enrolled mothers will be randomized to either the intervention (n=30; matched DHM) or control group (n=30; standard unmatched DHM). Infants of mothers assigned to the intervention group will receive "matched" DHM based on maternal secretor status, determined after randomization. Infant fecal samples will be collected weekly from soiled diapers until discontinuation of DHM or discharge/transfer from the unit. Samples of MOM and DHM will also be collected to analyze milk for HMO and nutrient content. Microbial DNA will be analyzed using 16S sequencing. Additionally, for a subset of samples selected based on 16S results, investigators will perform shotgun metagenomics to identify microbial population structures and functional capacity. Microbial composition from intervention (matched DHM), control (unmatched DHM) and reference (exclusive MOM) groups will be compared to determine differences in microbial diversity and taxonomy.

Impact on healthcare: If promising, investigators would like to examine this phenomenon in a much larger cohort of preterm infants from NICUs across Canada. This research could revolutionize how milk banks and neonatal intensive care units provide DHM to preterm infants. Finally, this research will expand on understanding of the prebiotic effects of HMOs on infant microbiome and may inform future prebiotic/probiotic supplementation regimens.

ELIGIBILITY:
Inclusion Criteria:

* Gestation up to 33 6/7 weeks at hospital admission (to guarantee at least 14 days intervention, since DHM fortification typically ends at 34+0 weeks adjusted gestational age).
* Provision of consent for infant to receive DHM.
* Mother has provided signed and dated informed consent and authorization to use protected health information, as required by national and local regulations.
* In the investigator's opinion, the subject mother understands and is able to comply with protocol requirements, instructions, and protocol-stated restrictions, and is likely to complete the study as planned.

Exclusion Criteria (Infant):

* Diagnosed with clinically significant major congenital malformation
* Intestinal perforation or stage 2 necrotizing enterocolitis (NEC)
* Unlikely to survive the study period
* Receiving extended courses of antibiotics (most infants are expected to receive up to 48hr antibiotic prophylaxis at birth according to standard NICU protocol; this criterion will only exclude infants receiving prolonged courses of antibiotics)
* Presence prior to enrollment of intestinal perforation or stage 2 necrotizing enterocolitis (NEC) prior to tolerating fortified feeds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fecal microbiome composition | sampled weekly until infant transferred from level III NICU, they are no longer receiving donor human milk or up to 60 days, whichever comes first.
  16S RNA sequencing of fecal bacteria

OTHER OUTCOMES:
Growth - weight | sampled weekly until infant transferred from level III NICU, they are no longer receiving donor human milk or up to 60 days, whichever comes first.
  measured in grams
Growth - length | sampled weekly until infant transferred from level III NICU, they are no longer receiving donor human milk or up to 60 days, whichever comes first.
  measured in centimetres
Growth - head circumference | sampled weekly until infant transferred from level III NICU, they are no longer receiving donor human milk or up to 60 days, whichever comes first.
  measured in centimetres
Days to full enteral feeds | Infant feeds are recorded daily, until infant transferred from level III NICU, they are no longer receiving donor human milk or up to 60 days, whichever comes first.
  Measure the number of days it takes from birth until the infant is taking 120 mL/kg/day (full feeds).
Length of Stay | Measured when infant is discharged or transferred from unit, or up to 60 days, whichever comes first.
  Time, measured in days, from admission (birth) to discharge or 'step-down' to level II NICU
Donor human milk composition - human milk oligosaccharide concentrations | Sampled from milk donations to the milk bank, up to 52 weeks postpartum
  Individual human milk oligosaccharides concentrations - measured in mol/mL
Donor human milk composition - nutritional composition | Sampled from milk donations to the milk bank, up to 52 weeks postpartum
  Micro-nutrients - measured in kcal/mL
Mothers own milk composition - Human milk oligosaccharide concentration | Sampled from one feeding of infant at 2 weeks post-birth.
  Human milk oligosaccharides concentrations - measured in mol/mL
Mothers own milk - nutritional composition | Sampled from one feeding of infant at 2 weeks post-birth.
  Micro-nutrients - measured in kcal/mL

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Azad, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
At this time we plan to share IPD within our research team only. We will consider sharing with other researchers in the future

REFERENCES:
- [Background] Azad MB, Robertson B, Atakora F, Becker AB, Subbarao P, Moraes TJ, Mandhane PJ, Turvey SE, Lefebvre DL, Sears MR, Bode L. Human Milk Oligosaccharide Concentrations Are Associated with Multiple Fixed and Modifiable Maternal Characteristics, Environmental Factors, and Feeding Practices. J Nutr. 2018 Nov 1;148(11):1733-1742. doi: 10.1093/jn/nxy175. PMID 30247646
- [Background] Bode L. Human milk oligosaccharides: every baby needs a sugar mama. Glycobiology. 2012 Sep;22(9):1147-62. doi: 10.1093/glycob/cws074. Epub 2012 Apr 18. PMID 22513036
- [Background] Marx C, Bridge R, Wolf AK, Rich W, Kim JH, Bode L. Human milk oligosaccharide composition differs between donor milk and mother's own milk in the NICU. J Hum Lact. 2014 Feb;30(1):54-61. doi: 10.1177/0890334413513923. Epub 2013 Nov 26. PMID 24282194
- [Background] Parra-Llorca A, Gormaz M, Alcantara C, Cernada M, Nunez-Ramiro A, Vento M, Collado MC. Preterm Gut Microbiome Depending on Feeding Type: Significance of Donor Human Milk. Front Microbiol. 2018 Jun 27;9:1376. doi: 10.3389/fmicb.2018.01376. eCollection 2018. PMID 29997594
- [Background] Lewis ZT, Totten SM, Smilowitz JT, Popovic M, Parker E, Lemay DG, Van Tassell ML, Miller MJ, Jin YS, German JB, Lebrilla CB, Mills DA. Maternal fucosyltransferase 2 status affects the gut bifidobacterial communities of breastfed infants. Microbiome. 2015 Apr 10;3:13. doi: 10.1186/s40168-015-0071-z. eCollection 2015. PMID 25922665
- See also: Lab Website — https://www.thrivediscovery.ca/